CLINICAL TRIAL: NCT04250337
Title: A Randomized, Double-Blind, Placebo-Controlled Trial To Evaluate The Efficacy and Safety of Lebrikizumab When Used In Combination With Topical Corticosteroid Treatment In Patients With Moderate-To-Severe Atopic Dermatitis
Brief Title: Safety and Efficacy of Lebrikizumab (LY3650150) in Combination With Topical Corticosteroid in Moderate-to-Severe Atopic Dermatitis.
Acronym: ADhere
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Dermira, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17803; 2019-004300-34 (EudraCT Number); J2T-DM-KGAD (Other: Eli Lilly and Company); DRM06-AD06 (Other: Dermira, Inc.)
Record Dates: First submitted 2020-01-30; First posted 2020-01-31 (Actual); Results first posted 2022-05-02 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Atopic Dermatitis
Keywords: Eczema; Dermatitis; Dermatitis, Atopic; Skin Diseases
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Dermatitis; Skin Diseases | interventions — lebrikizumab; Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, parallel group, placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lebrikizumab + Topical Corticosteroid (Experimental): 500 mg Lebrikizumab (2 x 250 mg) subcutaneous (SC) injections of lebrikizumab as a loading dose at Baseline and Week 2 followed by a single injection of 250 mg Lebrikizumab every 2 weeks (Q2W) from Week 4 until Week 14.
  Topical corticosteroid (TCS) will be initiated at Baseline in all participants and may be tapered or stopped, or restarted as needed, based on treatment response.
  Interventions: Biological: Lebrikizumab; Other: Topical Corticosteroid
- Placebo + Topical Corticosteroid (Placebo Comparator): Two placebo subcutaneous (SC) injections as a loading dose at Baseline and Week 2 followed by a single injection of placebo every Q2W from Week 4 until Week 14.
  TCS will be initiated at Baseline in all participants and may be tapered or stopped, or restarted as needed, based on treatment response
  Interventions: Other: Placebo; Other: Topical Corticosteroid

INTERVENTIONS:
Biological: Lebrikizumab — Subcutaneous injection
  Other Names: LY3650150; DRM06
  Arms: Lebrikizumab + Topical Corticosteroid
Other: Placebo — Subcutaneous injection
  Arms: Placebo + Topical Corticosteroid
Other: Topical Corticosteroid — Topical Corticosteroid

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel-group study which is 16 weeks in duration. The study is designed to evaluate the safety and efficacy of lebrikizumab when used in combination with topical corticosteroid (TCS) treatment compared with placebo in combination with TCS treatment for moderate-to-severe atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adult and adolescents (≥12 years to <18 years, and weighing ≥40 kg).
2. Chronic AD (according to American Academy of Dermatology Consensus Criteria) that has been present for ≥1 year before the screening visit.
3. Eczema Area and Severity Index (EASI) score ≥16 at the baseline visit.
4. Investigator Global Assessment (IGA) score ≥3 (scale of 0 to 4) at the baseline visit
5. ≥10% body surface area (BSA) of AD involvement at the baseline visit.
6. History of inadequate response to treatment with topical medications.

Exclusion Criteria:

1. Participation in a prior lebrikizumab clinical study.
2. Treatment with the following prior to the baseline visit:

   1. An investigational drug within 8 weeks or within 5 half-lives (if known), whichever is longer.
   2. Dupilumab within 8 weeks.
   3. B-cell-depleting biologics, including to rituximab, within 6 months.
   4. Other biologics within 5 half-lives (if known) or 16 weeks, whichever is longer.
3. Treatment with a live (attenuated) vaccine within 12 weeks of the baseline visit or planned during the study.
4. Uncontrolled chronic disease that might require bursts of oral corticosteroids.
5. Evidence of active acute or chronic hepatitis
6. History of human immunodeficiency virus (HIV) infection or positive HIV serology at screening.
7. History of malignancy, including mycosis fungoides, within 5 years before the screening visit, except completely treated in situ carcinoma of the cervix, completely treated and resolved non-metastatic squamous or basal cell carcinoma of the skin.
8. Pregnant or breastfeeding women, or women planning to become pregnant or breastfeed during the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2021-08-11 (Actual); Study Completion 2021-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (63):
- United States (43):
  - Investigate MD, Scottsdale, Arizona
  - Orange County Research Institute, Anaheim, California
  - Bakersfield Dermatology and Skin Cancer Medical Group, Bakersfield, California
  - Wallace Medical Group, Inc., Beverly Hills, California
  - First OC Dermatology, Fountain Valley, California
  - Center For Dermatology Clinical Research, Inc., Fremont, California
  - California Allergy and Asthma Medical Group + Research Center, Los Angeles, California
  - Keck School of Medicine University of Southern California, Los Angeles, California
  - Dermatology Research Associates, Los Angeles, California
  - LA Universal Research Center, INC, Los Angeles, California
  - ACRC Studies, San Diego, California
  - University Clinical Trials, Inc., San Diego, California
  - Southern California Dermatology, Inc., Santa Ana, California
  - Foxhall Dermatology, Washington D.C., District of Columbia
  - St. Francis Medical Institute, Clearwater, Florida
  - University of Florida - Gainesville, Gainesville, Florida
  - Direct Helpers Medical Center, Hialeah, Florida
  - The Community Research of South Florida, Hialeah, Florida
  - GSI Clinical Research, LLC, Margate, Florida
  - Vitae Research Center, LLC, Miami, Florida
  - Well Pharma Medical Research Corp., Miami, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Advanced Medical Research, Sandy Springs, Georgia
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - Dermatology and Skin Cancer Specialists, Rockville, Maryland
  - ActivMed Practices and Research, Beverly, Massachusetts
  - Beacon Clinical Research LLC, Quincy, Massachusetts
  - Fivenson Dermatology, Ann Arbor, Michigan
  - Clarkston Skin Research, Clarkston, Michigan
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - ALLCUTIS Research, Portsmouth, New Hampshire
  - Psoriasis Treatment Center of Central New Jersey, East Windsor, New Jersey
  - Sadick Research Group, New York, New York
  - OnSite Clinical Solutions, Charlotte, North Carolina
  - Wilmington Dermatology Center, Wilmington, North Carolina
  - Clinical Research Institute, Medford, Oregon
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Oregon Medical Research Center, Portland, Oregon
  - OHSU Center for Health and Healing, Portland, Oregon
  - Clinical Partners, LLC, Johnston, Rhode Island
  - Clinical Research Center of the Carolinas, Charleston, South Carolina
  - Arlington Research Center, Inc, Arlington, Texas
  - Dermatology Treatment and Research Center, Dallas, Texas
- Canada (6):
  - CARe Clinic, Red Deer, Alberta
  - Dr. Chih-ho Hong Medical Inc., Surrey, British Columbia
  - Enverus Medical Research, Surrey, British Columbia
  - Wiseman Dermatology Research Inc., Winnipeg, Manitoba
  - SKiN Centre for Dermatology, Peterborough, Ontario
  - International Dermatology Research, Montreal, Quebec
- Germany (5):
  - Klinikum der Johann Wolfgang Goethe-Universität Frankfurt, Frankfurt am Main, Hesse
  - Elbe Klinikum Buxtehude, Buxtehude, Lower Saxony
  - Technische Universitaet Dresden - Universitaetsklinikum Carl Gustav Carus - Klinik und Poliklinik fuer, Dresden, Saxony
  - Praxis für Ganzheitliche Dermatologie im Ärztehaus, Berlin
  - TFS Trial Form Support GmbH, Hamburg
- Poland (9):
  - DermMEDICA Sp. z o.o., Wroclaw, Lower Silesian Voivodeship
  - Alergo-Med Specjalistyczna Przychodnia Lekarska Sp Z O.O., Tarnów, Malopolska
  - Kliniczny Szpital Wojewodzki nr. 1 Klinika Dermatologii, Rzeszów, Podkarpackie Voivodeship
  - COPERNICUS Podmiot Leczniczy sp. z o.o., Gdansk, Pomeranian Voivodeship
  - Labderm s.c., Ossy, Silesian Voivodeship
  - Clinica Vitae Sp. z o.o., Gdansk, Woj. Pomorskie
  - Clinical Research Group Sp. z o.o., Warsaw
  - Centralny Szpital Kliniczny MSWiA, Warsaw
  - Gabinet Dermatlogiczny. Beata Krecisz, Kielce, Świętokrzyskie Voivodeship

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Simpson EL, Gooderham M, Wollenberg A, Weidinger S, Armstrong A, Soung J, Ferrucci S, Lima RG, Witte MM, Xu W, ElMaraghy H, Natalie CR, Pierce E, Blauvelt A; ADhere Investigators. Efficacy and Safety of Lebrikizumab in Combination With Topical Corticosteroids in Adolescents and Adults With Moderate-to-Severe Atopic Dermatitis: A Randomized Clinical Trial (ADhere). JAMA Dermatol. 2023 Feb 1;159(2):182-191. doi: 10.1001/jamadermatol.2022.5534. PMID 36630140
- See also: Safety and Efficacy of Lebrikizumab (LY3650150) in Combination With Topical Corticosteroid in Moderate-to-Severe Atopic Dermatitis. (ADhere) — https://trials.lillytrialguide.com/en-US/trial/4gJ6pg3ypXbcm8LEXb9M3b

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A participant is considered to have completed the study if he/she has completed the last scheduled visit:
  * For participants continuing into Long-term Extension (LTE), upon completion of week 16 visit and rolling into LTE study
  * For participants not continuing into LTE, when participant had either week 16 or Early Termination (ET) visit, and safety follow up visit (12 weeks after last study drug administration)
Groups:
- Placebo + Topical Corticosteroid: Two placebo subcutaneous (SC) injections as a loading dose at Baseline and Week 2 followed by a single injection of placebo every 2 weeks (Q2W) from Week 4 until Week 14.
  Topical Corticosteroid (TCS) will be initiated at Baseline in all participants and may be tapered or stopped, or restarted as needed, based on treatment response
- Lebrikizumab + Topical Corticosteroid: 500 milligram (mg) Lebrikizumab (2 x 250 mg) SC injections as a loading dose at Baseline and Week 2 followed by a single injection of 250 mg Lebrikizumab Q2W from Week 4 until Week 14.
  TCS will be initiated at Baseline in all participants and may be tapered or stopped, or restarted as needed, based on treatment response.
Period: Overall Study
Arm/Group | Placebo + Topical Corticosteroid | Lebrikizumab + Topical Corticosteroid
Started | 75 | 153
Received at Least One Dose of Study Drug | 75 | 153
Completed | 67 | 142
Not Completed | 8 | 11
Not completed — Adverse Event | 0 | 3
Not completed — Lack of Efficacy | 1 | 3
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Deviation | 2 | 2
Not completed — Withdrawal by Subject | 4 | 3

BASELINE CHARACTERISTICS:
Population: All randomized participants, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol.
Groups:
- Placebo + Topical Corticosteroid: Two placebo SC injections as a loading dose at Baseline and Week 2 followed by a single injection of placebo every Q2W from Week 4 until Week 14.
  TCS will be initiated at Baseline in all participants and may be tapered or stopped, or restarted as needed, based on treatment response.
- Lebrikizumab + Topical Corticosteroid: 500 mg Lebrikizumab (2 x 250 mg) SC injections of lebrikizumab as a loading dose at Baseline and Week 2 followed by a single injection of 250 mg Lebrikizumab Q2W from Week 4 until Week 14.
  TCS will be initiated at Baseline in all participants and may be tapered or stopped, or restarted as needed, based on treatment response
- Total: Total of all reporting groups
Arm/Group | Placebo + Topical Corticosteroid | Lebrikizumab + Topical Corticosteroid | Total
Number analyzed (Participants) | 75 | 153 | 228
Age, Customized [Count of Participants; unit: Participants]
  12 - <18 | 18 | 35 | 53
  >= 18 - <65 | 52 | 103 | 155
  >=65 - <75 | 5 | 10 | 15
  >=75 | 0 | 5 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 75 | 112
  Male | 38 | 78 | 116
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 5 | 7
  Asian | 13 | 18 | 31
  Native Hawaiian or Other Pacific Islander | 0 | 3 | 3
  Black or African American | 9 | 21 | 30
  White | 49 | 96 | 145
  More than one race | 1 | 8 | 9
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 8 | 14 | 22
  United States | 57 | 111 | 168
  Poland | 8 | 19 | 27
  Germany | 2 | 9 | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Investigator's Global Assessment (IGA) Score of 0 or 1 and a Reduction ≥2-points From Baseline to Week 16.
Description: The IGA measures the investigator's global assessment of the participant's overall severity of their AD, based on a static, numeric 5-point scale from 0 (clear skin) to 4 (severe disease). The score is based on an overall assessment of the degree of erythema, papulation/induration, oozing/crusting, and lichenification.
Time Frame: Baseline to Week 16
Population: All randomized participants, even if the participant did not take the assigned treatment, did not receive the correct treatment, or otherwise did not follow the protocol. One investigational site with seventeen participants was excluded from analysis due to Good Clinical Practice (GCP) issues.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo +Topical Corticosteroid: Two placebo SC injections as a loading dose at Baseline and Week 2 followed by a single injection of placebo Q2W from Week 4 until Week 14. TCS will be initiated at Baseline in all participants and may be tapered or stopped, or restarted as needed, based on treatment response.
- Lebrikizumab + Topical Corticosteroid: 500 mg Lebrikizumab (2 x 250 mg) SC injections as a loading dose at Baseline and Week 2 followed by a single injection 250 mg Lebrikizumab Q2W from Week 4 until Week 14.
  TCS will be initiated at Baseline in all participants and may be tapered or stopped, or restarted as needed, based on treatment response.
Arm/Group | Placebo +Topical Corticosteroid | Lebrikizumab + Topical Corticosteroid
Number analyzed (Participants) | 66 | 145
percentage of participants | 22.1 [11.6 to 32.7] | 41.2 [33.0 to 49.4]
Statistical Analysis 1: Comparison: Placebo +Topical Corticosteroid vs Lebrikizumab + Topical Corticosteroid; Test type: Superiority; p = 0.011, Cochran-Mantel-Haenszel; Risk Difference (RD) = 18.3, 95% CI 2-sided [5.1 to 31.5]

2. Primary Outcome: Percentage of Participants Achieving Eczema Area and Severity Index (EASI-75) (≥75% Reduction From Baseline in EASI Score) at Week 16
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe).
  The EASI responder is defined as a participant who achieves a ≥ 75% improvement from baseline in the EASI score.
Time Frame: Baseline to Week 16
Population: All randomized participants, even if the participant did not take the assigned treatment, did not receive the correct treatment, or otherwise did not follow the protocol. One investigational site with seventeen participants was excluded from analysis due to GCP issues.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo +Topical Corticosteroid | Lebrikizumab + Topical Corticosteroid
Number analyzed (Participants) | 66 | 145
percentage of participants | 42.2 [30.1 to 54.4] | 69.5 [61.9 to 77.2]
Statistical Analysis 1: Comparison: Placebo +Topical Corticosteroid vs Lebrikizumab + Topical Corticosteroid; Test type: Superiority; p < .001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 26.4, 95% CI 2-sided [12.1 to 40.8]

3. Secondary Outcome: Percentage of Participants Achieving EASI-90 (≥90% Reduction From Baseline in EASI Score) at Week 16
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe).
  The EASI responder is defined as a participant who achieves a ≥ 90% improvement from baseline in the EASI score.
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo +Topical Corticosteroid | Lebrikizumab + Topical Corticosteroid
Number analyzed (Participants) | 66 | 145
percentage of participants | 21.7 [11.4 to 32.0] | 41.2 [33.0 to 49.3]
Statistical Analysis 1: Comparison: Placebo +Topical Corticosteroid vs Lebrikizumab + Topical Corticosteroid; Test type: Superiority; p = 0.008, Cochran-Mantel-Haenszel; Risk Difference (RD) = 18.9, 95% CI 2-sided [6.1 to 31.7]

4. Secondary Outcome: Percent Change in Pruritus Numerical Rating Scale (NRS) Score From Baseline to Week 16
Description: Pruritus NRS is an 11-point scale used by participants to rate their worst itch severity over the past 24 hours with 0 indicating "No itch" and 10 indicating "Worst itch imaginable." Least Squares (LS) Mean was calculated using analysis covariance (ANCOVA) model includes treatment, baseline value, and stratification factors of geographic region, age group, baseline IGA score as fixed factors.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo +Topical Corticosteroid | Lebrikizumab + Topical Corticosteroid
Number analyzed (Participants) | 63 | 139
Percent change | -35.47 (6.358) | -50.68 (4.546)
Statistical Analysis 1: Comparison: Placebo +Topical Corticosteroid vs Lebrikizumab + Topical Corticosteroid; Test type: Superiority; p = 0.017263, ANCOVA; LS Mean Difference (Final Values) = -15.21, 95% CI 2-sided [-27.7 to -2.7], Standard Error of Mean 6.373

5. Secondary Outcome: Percentage of Participants With a Pruritus NRS of ≥4-Points at Baseline Who Achieve a ≥4-Point Reduction From Baseline to Week 16
Description: Pruritus NRS is an 11-point scale used by participants to rate their worst itch severity over the past 24 hours with 0 indicating "No itch" and 10 indicating "Worst itch imaginable."
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo +Topical Corticosteroid | Lebrikizumab + Topical Corticosteroid
Number analyzed (Participants) | 57 | 130
percentage of participants | 31.9 [19.3 to 44.4] | 50.6 [41.8 to 59.4]
Statistical Analysis 1: Comparison: Placebo +Topical Corticosteroid vs Lebrikizumab + Topical Corticosteroid; Test type: Superiority; p = 0.017, Cochran-Mantel-Haenszel; Risk Difference (RD) = 19.2, 95% CI 2-sided [4.3 to 34.1]

6. Secondary Outcome: Percentage of Participants With a Pruritus NRS of ≥5-points at Baseline Who Achieve a ≥4-point Reduction From Baseline to Week 16
Description: as for outcome 5
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo +Topical Corticosteroid | Lebrikizumab + Topical Corticosteroid
Number analyzed (Participants) | 53 | 124
percentage of participants | 26.4 [14.5 to 38.3] | 46.8 [38.0 to 55.6]
Statistical Analysis 1: Comparison: Placebo +Topical Corticosteroid vs Lebrikizumab + Topical Corticosteroid; Test type: Superiority; p = 0.007, Cochran-Mantel-Haenszel; Risk Difference (RD) = 21.6, 95% CI 2-sided [7.1 to 36.1]

7. Secondary Outcome: Percent Change in EASI Score From Baseline at Week 16
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe).
  LS Mean was calculated using ANCOVA model with treatment, baseline value, and stratification factors of geographic region, age group, baseline IGA score (IGA 3 versus 4) as fixed factors.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo +Topical Corticosteroid | Lebrikizumab + Topical Corticosteroid
Number analyzed (Participants) | 66 | 145
Percent Change | -53.12 (5.097) | -76.76 (4.119)
Statistical Analysis 1: Comparison: Placebo +Topical Corticosteroid vs Lebrikizumab + Topical Corticosteroid; Test type: Superiority; p = 0.000003, ANCOVA; LS Mean Difference (Final Values) = -23.64, 95% CI 2-sided [-33.6 to -13.7], Standard Error of Mean 5.074

8. Secondary Outcome: Change From Baseline to Week 16 in Percent Body Surface Area (BSA)
Description: The BSA affected by AD will be assessed for 4 separate body regions: head and neck, trunk (including genital region), upper extremities, and lower extremities (including the buttocks). Each body region will be assessed for disease extent ranging from 0% to 100% involvement. BSA was calculated using the participant's palm using the 1% rule, 1 palm was equivalent to 1% with estimates of the number of palms it takes to cover the affected AD area. Maximum number of palms were 10 palms for head and neck (10%), 20 palms for upper extremities (20%), 30 palms for trunk, including axilla and groin (30%), 40 palms for lower extremities, including buttocks (40%). Percent of BSA for a body region was calculated as = total number of palms in a body region * % surface area equivalent to 1 palm. Overall percent BSA of all 4 body regions ranges from 0% to 100 % with higher values representing greater severity of AD.
Time Frame: Baseline, Week 16
Population: All randomized participants, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. The mixed model repeated measure (MMRM) include treatment, visit, the interaction of treatment by-visit, geographic region, age group, baseline IGA score. One investigational site with seventeen participants was excluded from analysis due to GCP issues.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo +Topical Corticosteroid | Lebrikizumab + Topical Corticosteroid
Number analyzed (Participants) | 53 | 130
score on a scale | 16.92 (2.287) | -29.19 (1.686)
Statistical Analysis 1: Comparison: Placebo +Topical Corticosteroid vs Lebrikizumab + Topical Corticosteroid; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference (Final Values) = -12.28, 95% CI 2-sided [-17.07 to -7.49], Standard Error of Mean 2.428

9. Secondary Outcome: Percentage of Participants Achieving EASI-90 at Week 4
Description: as for outcome 3
Time Frame: Baseline to Week 4
Population: All randomized participants, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. One investigational site with seventeen participants was excluded from analysis due to GCP issues.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo +Topical Corticosteroid | Lebrikizumab + Topical Corticosteroid
Number analyzed (Participants) | 66 | 145
percentage of participants | 7.2 [0.5 to 13.8] | 10.7 [5.6 to 15.8]
Statistical Analysis 1: Comparison: Placebo +Topical Corticosteroid vs Lebrikizumab + Topical Corticosteroid; Test type: Superiority; p = 0.454, Cochran-Mantel-Haenszel; Risk Difference (RD) = 3.5, 95% CI 2-sided [-4.9 to 11.8]

10. Secondary Outcome: Percent Change in Sleep-loss Score From Baseline to Week 16
Description: Sleep Loss due to interference of itch will be assessed by the participant. Participants rate their interference of itch on sleep based on a 5-point Likert scale [0 (not at all) to 4 (unable to sleep at all)]. Higher scores indicated a greater impact and worse outcome. Assessments will be recorded daily by the participant using an electronic diary. LS Mean was calculated using ANCOVA model with treatment, baseline value, and stratification factors of geographic region, age group, baseline IGA (3 versus 4) score as fixed factors.
  .
Time Frame: Baseline, Week 16
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo +Topical Corticosteroid | Lebrikizumab + Topical Corticosteroid
Number analyzed (Participants) | 62 | 134
percent change | -36.89 (12.217) | -57.03 (7.939)
Statistical Analysis 1: Comparison: Placebo +Topical Corticosteroid vs Lebrikizumab + Topical Corticosteroid; Test type: Superiority; p = 0.117607, ANCOVA; Markov Chain Monte Carlo (MCMC) = -20.14, 95% CI 2-sided [-45.4 to 5.1], Standard Error of Mean 12.810

11. Secondary Outcome: Change From Baseline in Sleep-loss Score at Week 16
Description: Sleep Loss due to interference of itch will be assessed by the participant. Participants rate their interference of itch on sleep based on a 5-point Likert scale [0 (not at all) to 4 (unable to sleep at all)]. Higher scores indicated a greater impact and worse outcome. Assessments will be recorded daily by the participant using an electronic diary. LS Mean was calculated using ANCOVA model with treatment, baseline value, and stratification factors of geographic region, age group, baseline IGA (3 versus 4) score as fixed factors.
  APD: All randomized participants, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol.
Time Frame: Baseline, Week 16
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo +Topical Corticosteroid | Lebrikizumab + Topical Corticosteroid
Number analyzed (Participants) | 63 | 139
score on a scale | -0.80 (0.132) | -1.10 (0.102)
Statistical Analysis 1: Comparison: Placebo +Topical Corticosteroid vs Lebrikizumab + Topical Corticosteroid; Test type: Superiority; p = 0.025293, ANCOVA; Markov Chain Monte Carlo (MCMC) = -0.30, 95% CI 2-sided [-0.6 to -0.0], Standard Error of Mean 0.134

12. Secondary Outcome: Percentage of Participants With a Pruritus NRS of ≥4-points at Baseline Who Achieve a ≥4-point Reduction From Baseline to Week 4
Description: The Pruritus NRS is an 11-point scale used by participants to assess their worst itch severity over the past 24 hours, with 0 indicating no itch and 10 indicating worst itch imaginable.
Time Frame: Baseline to Week 4
Population: All randomized participants, with baseline Pruritus NRS score of at least 4, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. One investigational site with seventeen participants was excluded from analysis due to GCP issues.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo +Topical Corticosteroid | Lebrikizumab + Topical Corticosteroid
Number analyzed (Participants) | 57 | 130
percentage of participants | 9.3 [1.6 to 17.1] | 23.5 [16.2 to 30.9]
Statistical Analysis 1: Comparison: Placebo +Topical Corticosteroid vs Lebrikizumab + Topical Corticosteroid; Test type: Superiority; p = 0.022, Cochran-Mantel-Haenszel; Risk Difference (RD) = 14.2, 95% CI 2-sided [3.8 to 24.7]

13. Secondary Outcome: Percentage of Participants With a Pruritus NRS of ≥4-points at Baseline Who Achieve a ≥4-point Reduction From Baseline to Week 2
Description: as for outcome 12
Time Frame: Baseline to Week 2
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo +Topical Corticosteroid: Two placebo SC injections as a loading dose at Baseline and Week 2 followed by a single injection of placebo Q2W from Week 4 until Week 14.TCS will be initiated at Baseline in all participants and may be tapered or stopped, or restarted as needed, based on treatment response.
Arm/Group | Placebo +Topical Corticosteroid | Lebrikizumab + Topical Corticosteroid
Number analyzed (Participants) | 57 | 130
percentage of participants | 7.1 [0.4 to 13.8] | 8.5 [3.7 to 13.3]
Statistical Analysis 1: Comparison: Placebo +Topical Corticosteroid vs Lebrikizumab + Topical Corticosteroid; Test type: Superiority; p = 0.764, Cochran-Mantel-Haenszel; Risk Difference (RD) = 1.2, 95% CI 2-sided [-7.3 to 9.7]

14. Secondary Outcome: Percentage of Participants With a Pruritus NRS of ≥4-points at Baseline Who Achieve a ≥4-point Reduction From Baseline to Week 1
Description: as for outcome 12
Time Frame: Baseline to Week 1
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo +Topical Corticosteroid | Lebrikizumab + Topical Corticosteroid
Number analyzed (Participants) | 57 | 130
percentage of participants | 1.8 [0.0 to 5.2] | 3.8 [0.5 to 7.2]
Statistical Analysis 1: Comparison: Placebo +Topical Corticosteroid vs Lebrikizumab + Topical Corticosteroid; Test type: Superiority; p = 0.498, Cochran-Mantel-Haenszel; Risk Difference (RD) = 1.9, 95% CI 2-sided [-2.9 to 6.7]

15. Secondary Outcome: Percentage of Participants With a Pruritus NRS of ≥5-points at Baseline Who Achieve a ≥4-point Reduction From Baseline to Week 4
Description: as for outcome 12
Time Frame: Baseline to Week 4
Population: All randomized participants, with baseline Pruritus NRS score of at least 5, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. One investigational site with seventeen participants was excluded from analysis due to GCP issues.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo +Topical Corticosteroid | Lebrikizumab + Topical Corticosteroid
Number analyzed (Participants) | 53 | 124
percentage of participants | 7.5 [0.4 to 14.7] | 23.4 [15.9 to 30.8]
Statistical Analysis 1: Comparison: Placebo +Topical Corticosteroid vs Lebrikizumab + Topical Corticosteroid; Test type: Superiority; p = 0.014, Cochran-Mantel-Haenszel; Risk Difference (RD) = 15.6, 95% CI 2-sided [5.3 to 25.9]

16. Secondary Outcome: Percentage of Participants With a Pruritus NRS of ≥5-points at Baseline Who Achieve a ≥4-point Reduction From Baseline to Week 2
Description: as for outcome 12
Time Frame: Baseline to Week 2
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo +Topical Corticosteroid | Lebrikizumab + Topical Corticosteroid
Number analyzed (Participants) | 53 | 124
percentage of participants | 7.5 [0.4 to 14.7] | 8.9 [3.9 to 13.9]
Statistical Analysis 1: Comparison: Placebo +Topical Corticosteroid vs Lebrikizumab + Topical Corticosteroid; Test type: Superiority; p = 0.818, Cochran-Mantel-Haenszel; Risk Difference (RD) = 1.1, 95% CI 2-sided [-8.0 to 10.2]

17. Secondary Outcome: Percentage of Participants With a Pruritus NRS of ≥5-points at Baseline Who Achieve a ≥4-point Reduction From Baseline to Week 1
Description: as for outcome 12
Time Frame: Baseline to Week 1
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo +Topical Corticosteroid | Lebrikizumab + Topical Corticosteroid
Number analyzed (Participants) | 53 | 124
percentage of participants | 1.9 [0.0 to 5.5] | 4.0 [0.6 to 7.5]
Statistical Analysis 1: Comparison: Placebo +Topical Corticosteroid vs Lebrikizumab + Topical Corticosteroid; Test type: Superiority; p = 0.499, Cochran-Mantel-Haenszel; Risk Difference (RD) = 2.0, 95% CI 2-sided [-3.1 to 7.1]

18. Secondary Outcome: Percentage of Topical Corticosteroid (TCS)/Topical Calcineurin Inhibitors (TCI) Free Days From Baseline to Week 16
Description: Number of the total TCS/TCI free days divided by total number of days during the treatment period. The mixed model repeated measures (MMRM) includes treatment, visit, the interaction of treatment by-visit, geographic region, age group, baseline IGA score.
Time Frame: Baseline to Week 16
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: Percentage of Days
Arm/Group | Placebo +Topical Corticosteroid | Lebrikizumab + Topical Corticosteroid
Number analyzed (Participants) | 53 | 131
Percentage of Days | 23.88 (4.823) | 31.17 (3.512)
Statistical Analysis 1: Comparison: Placebo +Topical Corticosteroid vs Lebrikizumab + Topical Corticosteroid; Test type: Superiority; p = 0.155, Mixed Models Analysis; LS Mean Difference (Final Values) = 7.29, 95% CI 2-sided [-2.78 to 17.36], Standard Error of Mean 5.104

19. Secondary Outcome: Median Time (Days) to TCS/TCI-free Use From Baseline to Week 16
Description: Days from first study drug injection to the day participant stopped using all TCS/TCI (if a participant started and stopped using low or midpotency TCS/TCI multiple times, use the last stop date as the stop date for this participant).
Time Frame: Baseline to Week 16
Population: as for outcome 9
Measure: Median (Full Range); unit: days
Arm/Group | Placebo +Topical Corticosteroid | Lebrikizumab + Topical Corticosteroid
Number analyzed (Participants) | 66 | 145
days | NA [1 to 112] — Less than 50 % of the participants reached TCS free within treatment window, median was not calculable. | 121.0 [2 to 121]

20. Secondary Outcome: Percent Change in SCORing Atopic Dermatitis (SCORAD) From Baseline to Week 16
Description: The SCORAD index uses the rule of nines to assess disease extent and evaluates 6 clinical characteristics to determine disease severity: (1) erythema, (2) edema/papulation, (3) oozing/crusts, (4) excoriation, (5) lichenification, and (6) dryness on a scale of 0 to 3 (0=absence, 1=mild, 2=moderate, 3=severe). The SCORAD index also assesses subjective symptoms of pruritus and sleep loss with VAS where 0 is no itching or no trouble sleeping and 10 is unbearable itching or a lot of trouble sleeping. These 3 aspects: extent of disease (A: 0-1-2), disease severity (B: 0-18), & subjective symptoms (C: 0-20) combine using A/5 + 7*B/2+ C to give a maximum possible score of 103, where 0 = no disease and 103 = severe disease.
  LS Mean was calculated using the ANCOVA model with treatment group, baseline value, and stratification factors of geographic region, age group, baseline IGA (3 versus 4) score as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. One investigational site with seventeen participants was excluded from analysis due to GCP issues. Missing Values were imputed using last observation carried forward (LOCF) method.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo +Topical Corticosteroid | Lebrikizumab + Topical Corticosteroid
Number analyzed (Participants) | 65 | 140
percent change | -37.35 (4.415) | -55.04 (3.542)
Statistical Analysis 1: Comparison: Placebo +Topical Corticosteroid vs Lebrikizumab + Topical Corticosteroid; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference (Final Values) = -17.69, 95% CI 2-sided [-26.37 to -9.01], Standard Error of Mean 4.403

21. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) at Week 16
Description: The DLQI is a 10-item, validated questionnaire used to assess the impact of skin disease on the quality of life of an affected person. The 10 questions cover the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, and treatment, over the previous week. Response categories include "Not at all," "A little," "A lot," and "Very much," with corresponding scores of 0, 1, 2, and 3 respectively. Questions 3-10 also have an additional response category of "Not relevant" which is scored as "0". Questions are scored from 0 to 3, giving a possible total score range from 0 (no impact of skin disease on quality of life) to 30 (maximum impact on quality of life). A high score is indicative of a poor quality of life.
  LS Mean was calculated using the ANCOVA model with treatment, baseline value, and stratification factors of geographic region, age group, baseline IGA (3 versus 4) score as fixed factors.
Time Frame: Baseline, Week 16
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo +Topical Corticosteroid | Lebrikizumab + Topical Corticosteroid
Number analyzed (Participants) | 51 | 109
score on a scale | -6.46 (1.855) | -9.79 (1.815)
Statistical Analysis 1: Comparison: Placebo +Topical Corticosteroid vs Lebrikizumab + Topical Corticosteroid; Test type: Superiority; p = 0.001031, ANCOVA; LS Mean Difference (Final Values) = -3.33, 95% CI 2-sided [-5.3 to -1.3], Standard Error of Mean 1.014

22. Secondary Outcome: Percentage of Participants With a DLQI Score ≥4 Points at Baseline Who Achieve a ≥4 Points
Description: as for outcome 21
Time Frame: Baseline to Week 16
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo +Topical Corticosteroid | Lebrikizumab + Topical Corticosteroid
Number analyzed (Participants) | 48 | 105
percentage of participants | 58.7 [44.1 to 73.2] | 77.4 [69.3 to 85.5]
Statistical Analysis 1: Comparison: Placebo +Topical Corticosteroid vs Lebrikizumab + Topical Corticosteroid; Test type: Superiority; p = 0.036, Cochran-Mantel-Haenszel; Risk Difference (RD) = 17.2, 95% CI 2-sided [0.1 to 34.3]

23. Secondary Outcome: Change From Baseline in European Quality of Life-5 Dimensions (EQ-5D) at Week 16 Health State Index
Description: The EQ-5D-5L is a 2-part measurement. The first part is comprised of the following 5 participant-reported dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The responses are used to derive the health state index scores using the United Kingdom (UK) algorithm, with scores ranging from -0.594 to 1, and the United States (US) algorithm, with scores ranging from -0.109 to 1, with higher score indicating better health state.
  LS Mean was calculated using the ANCOVA model with treatment, baseline value, and stratification factors of geographic region, age group, baseline IGA (3 versus 4) score as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. One investigational site with seventeen participants was excluded from analysis due to GCP issues. Missing values were imputed using LOCF method.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo +Topical Corticosteroid | Lebrikizumab + Topical Corticosteroid
Number analyzed (Participants) | 66 | 143
score on a scale
  Health State Index UK | 0.05 (0.025) | 0.15 (0.019)
  Health State Index US | 0.03 (0.018) | 0.10 (0.014)
Statistical Analysis 1: Comparison: Placebo +Topical Corticosteroid vs Lebrikizumab + Topical Corticosteroid; Health State Index UK; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference (Final Values) = 0.11, 95% CI 2-sided [0.06 to 0.16], Standard Error of Mean 0.025
Statistical Analysis 2: Comparison: Placebo +Topical Corticosteroid vs Lebrikizumab + Topical Corticosteroid; Health State Index US; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference (Final Values) = 0.07, 95% CI 2-sided [0.04 to 0.11], Standard Error of Mean 0.018

24. Secondary Outcome: Change From Baseline in European Quality of Life-5 Dimensions (EQ-5D) at Week 16 Visual Analog Score (VAS)
Description: The EQ-5D-5L is a 2-part measurement. The second part is assessed using a VAS that ranged from 0 to 100 millimeter (mm), where 0 is the worst health you can imagine and 100 is the best health you can imagine. LS Mean was calculated using the ANCOVA model with treatment, baseline value, and stratification factors of geographic region, age group, baseline IGA (3 versus 4) score as fixed factors.
Time Frame: Baseline, Week 16
Population: as for outcome 23
Measure: Least Squares Mean (Standard Error); unit: millimeters (mm)
Arm/Group | Placebo +Topical Corticosteroid | Lebrikizumab + Topical Corticosteroid
Number analyzed (Participants) | 65 | 143
millimeters (mm) | 6.51 (2.364) | 10.13 (1.831)
Statistical Analysis 1: Comparison: Placebo +Topical Corticosteroid vs Lebrikizumab + Topical Corticosteroid; Test type: Superiority; p = 0.131, ANCOVA; LS Mean Difference (Final Values) = 3.62, 95% CI 2-sided [-1.08 to 8.32], Standard Error of Mean 2.386

25. Secondary Outcome: Change From Baseline in Patient Oriented Eczema Measure (POEM) at Week 16
Description: POEM is a 7-item, validated, questionnaire used by the participant to assess disease symptoms over the last week. The participant is asked to respond to 7 questions on skin dryness, itching, flaking, cracking, sleep loss, bleeding and weeping. All 7 answers carry equal weight with a total possible score from 0 to 28 (answers scored as: No days=0; 1- 2 days = 1; 3-4 days = 2; 5-6 days = 3; everyday = 4). A high score is indicative of a poor quality of life. POEM responses will be captured using an electronic diary and transferred into the clinical database. LS Mean was calculated using MMRM model using treatment, baseline value, visit, the interaction of the baseline value-by-visit, the interaction of treatment by-visit as covariates, geographic region, age group, baseline IGA (3 versus 4) score as fixed.
Time Frame: Baseline, Week 16
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo +Topical Corticosteroid | Lebrikizumab + Topical Corticosteroid
Number analyzed (Participants) | 40 | 101
score on a scale | -6.24 (1.038) | -10.23 (0.727)
Statistical Analysis 1: Comparison: Placebo +Topical Corticosteroid; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference (Final Values) = -4.00, 95% CI 2-sided [-6.26 to -1.74], Standard Error of Mean 1.145

26. Secondary Outcome: Change From Baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety at Week 16 - Adults
Description: PROMIS is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. The PROMIS measures will be completed by the participant in the study clinic. PROMIS anxiety has 8 questions on Emotion Distress-Anxiety. Each question has 5 response options with values from 1 to 5. Total raw scores were converted to T-scores with higher scores indicating greater severity of symptoms. LS Mean was calculated using the ANCOVA model with treatment, baseline value, and stratification factors of geographic region, age group, baseline IGA (3 versus 4) score as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. One investigational site with seventeen participants was excluded from analysis due to GCP issues. Missing values were imputed with the LOCF method.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo +Topical Corticosteroid | Lebrikizumab + Topical Corticosteroid
Number analyzed (Participants) | 43 | 101
score on a scale | -1.08 (1.367) | -1.88 (1.027)
Statistical Analysis 1: Comparison: Placebo +Topical Corticosteroid vs Lebrikizumab + Topical Corticosteroid; Test type: Superiority; p = 0.571, ANCOVA; LS Mean Difference (Final Values) = -0.80, 95% CI 2-sided [-3.58 to 1.98], Standard Error of Mean 1.407

27. Secondary Outcome: Change From Baseline in PROMIS Depression at Week 16 - Adults
Description: PROMIS is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. The PROMIS measures will be completed by the participant in the study clinic. PROMIS depression has 8 questions on Emotion Distress-Depression. Each question has 5 response options with values from 1 to 5. Total raw scores were converted to T-scores with higher scores indicating greater severity of symptoms. LS Mean was calculated using the ANCOVA model with treatment, baseline value, and stratification factors of geographic region, age group, baseline IGA (3 versus 4) score as fixed factors.
Time Frame: Baseline, Week 16
Population: as for outcome 26
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo +Topical Corticosteroid | Lebrikizumab + Topical Corticosteroid
Number analyzed (Participants) | 43 | 101
score on a scale | -1.21 (1.098) | -1.38 (0.834)
Statistical Analysis 1: Comparison: Placebo +Topical Corticosteroid vs Lebrikizumab + Topical Corticosteroid; Test type: Superiority; p = 0.882, ANCOVA; LS Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-2.40 to 2.06], Standard Error of Mean 1.127

28. Secondary Outcome: Change From Baseline in PROMIS Anxiety at Week 16 - Pediatrics
Description: PROMIS® is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. Participants ≤17 years will complete pediatric versions for the duration of the study. PROMIS anxiety has 8 questions on Emotion Distress-Anxiety (or Pediatric Anxiety Symptom). Each question has 5 response options with values from 1 to 5. Total raw scores were converted to T-scores with higher scores indicating greater severity of symptoms. LS Mean was calculated using the ANCOVA model with treatment, baseline value, and stratification factors of geographic region, age group, baseline IGA (3 versus 4) score as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. One investigational site with seventeen participants was excluded from analysis due to GCP issues. Missing values were imputed using the LOCF method.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo +Topical Corticosteroid | Lebrikizumab + Topical Corticosteroid
Number analyzed (Participants) | 13 | 31
score on a scale | -4.92 (2.333) | -1.46 (1.732)
Statistical Analysis 1: Comparison: Placebo +Topical Corticosteroid vs Lebrikizumab + Topical Corticosteroid; Test type: Superiority; p = 0.171, ANCOVA; LS Mean Difference (Final Values) = 3.46, 95% CI 2-sided [-1.56 to 8.48], Standard Error of Mean 2.480

29. Secondary Outcome: Change From Baseline in PROMIS Depression at Week 16 - Pediatrics
Description: PROMIS® is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. Participants ≤17 years will complete pediatric versions for the duration of the study. PROMIS depression has 8 questions on Emotion Distress-Depression (or Pediatric Depressive Symptom). Each question has 5 response options with values from 1 to 5. Total raw scores were converted to T-scores with higher scores indicating greater severity of symptoms. LS Mean was calculated using the ANCOVA model with treatment, baseline value, and stratification factors of geographic region, age group, baseline IGA (3 versus 4) score as fixed factors.
Time Frame: Baseline, Week 16
Population: as for outcome 28
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo +Topical Corticosteroid | Lebrikizumab + Topical Corticosteroid
Number analyzed (Participants) | 13 | 31
score on a scale | -6.43 (2.536) | -2.01 (1.916)
Statistical Analysis 1: Comparison: Placebo +Topical Corticosteroid vs Lebrikizumab + Topical Corticosteroid; Test type: Superiority; p = 0.109, ANCOVA; LS Mean Difference (Final Values) = 4.43, 95% CI 2-sided [-1.03 to 9.89], Standard Error of Mean 2.697

30. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire (ACQ-5) Score at Week 16 in Participants Who Have Self-reported Comorbid Asthma
Description: The ACQ-5 has been shown to reliably measure asthma control and distinguish participants with well-controlled asthma (score ≤0.75 points) from those with uncontrolled asthma (score ≥1.5 points). It consists of 5 questions that are scored on a 7- point Likert scale with a recall period of 1 week. The total ACQ-5 score is the mean score of all questions; a lower score represents better asthma control.
  LS Mean was calculated using ANCOVA with treatment, baseline value, geographic region, age group, baseline IGA (3 versus 4) score as fixed factors.
Time Frame: Baseline, Week 16
Population: as for outcome 26
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo +Topical Corticosteroid | Lebrikizumab + Topical Corticosteroid
Number analyzed (Participants) | 14 | 38
score on a scale | 0.12 (0.116) | 0.13 (0.076)
Statistical Analysis 1: Comparison: Placebo +Topical Corticosteroid vs Lebrikizumab + Topical Corticosteroid; Test type: Superiority; p = 0.922, ANCOVA; LS Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.22 to 0.24], Standard Error of Mean 0.116

31. Secondary Outcome: Change From Baseline in Children's Dermatology Life Quality Index (CDLQI) at Week 16
Description: The CDLQI questionnaire is designed for use in children (4 to 16 years of age). It consists of 10 items that are grouped into 6 domains: symptoms & feelings, leisure, school or holidays, personal relationships, sleep, & treatment. The scoring of each question is: Very much =3; Quite a lot = 2; Only a little = 1; Not at all = 0. CDLQI total score is calculated by summing all 10 items responses, and has a range of 0 to 30 (higher scores are indicative of greater impairment).
  LS Mean was calculated using MMRM model which includes treatment, baseline value, visit, the interaction of the baseline value-by-visit as covariates, the interaction of treatment by-visit, geographic region, age group, and baseline IGA (3 versus 4) score as fixed factors.
Time Frame: Baseline, Week 16
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo +Topical Corticosteroid | Lebrikizumab + Topical Corticosteroid
Number analyzed (Participants) | 11 | 24
score on a scale | -4.71 (1.170) | -9.33 (0.887)
Statistical Analysis 1: Comparison: Placebo +Topical Corticosteroid vs Lebrikizumab + Topical Corticosteroid; Test type: Superiority; p = 0.001, Mixed Models Analysis; LS Mean Difference (Final Values) = -4.62, 95% CI 2-sided [-7.22 to -2.03], Standard Error of Mean 1.271

ADVERSE EVENTS:
Time Frame: Baseline up to Week 28
Description: All randomized participants who received at least 1 dose of study treatment.
Groups:
- Placebo +Topical Corticosteroid: Two placebo SC injections as a loading dose at Baseline and Week 2 followed by a single injection of placebo Q2W from Week 4 until Week 14. Topical corticosteroid (TCS) will be initiated at Baseline in all participants and may be tapered or stopped, or restarted as needed, based on treatment response.
- Lebrikizumab + Topical Corticosteroid: 500 mg Lebrikizumab (2 x 250 mg) subcutaneous (SC) injections as a loading dose at Baseline and Week 2 followed by a single injection of 250 mg Lebrikizumab every 2 weeks (Q2W) from Week 4 until Week 14. Topical corticosteroid (TCS) will be initiated at Baseline in all participants and may be tapered or stopped, or restarted as needed, based on treatment response.
Arm/Group | Placebo +Topical Corticosteroid | Lebrikizumab + Topical Corticosteroid
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/153
Serious Adverse Events (participants affected / at risk) | 1/75 | 2/153
Other Adverse Events (participants affected / at risk) | 26/75 | 66/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo +Topical Corticosteroid (N=75) | Lebrikizumab + Topical Corticosteroid (N=153)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo +Topical Corticosteroid (N=75) | Lebrikizumab + Topical Corticosteroid (N=153)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Lymphocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Blepharitis (Eye disorders) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 3 (3)
Eye irritation (Eye disorders) | 0 (0) | 1 (2)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1)
Vernal keratoconjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Xerophthalmia (Eye disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Injection site erythema (General disorders) | 0 (0) | 1 (1)
Injection site pruritus (General disorders) | 0 (0) | 1 (2)
Injection site rash (General disorders) | 0 (0) | 2 (2)
Injection site reaction (General disorders) | 1 (1) | 2 (2)
Injection site swelling (General disorders) | 0 (0) | 1 (1)
Vaccination site pain (General disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Bacterial colitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 7 (8)
Covid-19 (Infections and infestations) | 0 (0) | 2 (2)
Furuncle (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 2 (2)
Impetigo (Infections and infestations) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 5 (6) | 3 (5)
Ophthalmic herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 2 (2)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Suture related complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 1 (2)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1)
Weight increased (Investigations) | 0 (0) | 1 (1)
Alcohol intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Vitamin d deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 7 (7)
Ophthalmic migraine (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Alopecia areata (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin lesion inflammation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Hypertension (Vascular disorders) | 1 (1) | 4 (4)

LIMITATIONS AND CAVEATS:
One investigational site with seventeen participants was excluded from analysis due to GCP issues.

Because of an error in the electronic data collection tool, the actual maximum score for each of the SCORAD symptoms was 9 instead of 10, resulting in a total maximum SCORAD score of 101 instead of 103. During the study, discussions with the SCORAD copyright owner resulted in a decision not to adjust the scale used or notify investigators as the altered scale was not expected to bias the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-05-13): https://cdn.clinicaltrials.gov/large-docs/37/NCT04250337/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/37/NCT04250337/SAP_001.pdf